CLINICAL TRIAL: NCT02001805
Title: Fitness, Glucosemetabolism, Cognitive Function, Bodycomposition and Muscular Function in Active Runners and Matched Controls
Brief Title: Marathon Runners Compared to Sedentary Matched Control Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inge Holm (Other)
Collaborators: The Augustinus Foundation, Denmark. (Other)
Responsible Party: Sponsor-Investigator, Inge Holm, Head of Section CIM, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: Marathon Cohorte
Record Dates: First submitted 2011-05-18; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma, muscle tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Marathon runners: Very active runners that have been running > 10 marathons, 2 within the last year, or an amount of 50 km/week for the last 5 years
- Control subjects: Healthy normal weight control subjects, with a low activity level < 1 hour phsyical activity pr. week. They are matched with runners on age, BMI and gender

SUMMARY:
The investigators wish to compare very active runners in healthy untrained control subjects on a number of parameters.

The project aims to understand the underlying mechanisms by which physical inactivity causes diseases. This the investigators will study the full spectrum of physical activity, from the most inert of the most active people. The investigators have already collected muscle biopsies and established stem cells from people with Type 2 diabetes, obese healthy and normal weight healthy. In this study, the investigators will establish a cohort of highly physically active marathon runners. In a case-control design, the investigators compare muscle stem cell function across the entire spectrum of physical activity / inactivity.

DETAILED DESCRIPTION:
There has never been as much focus on running as in these days. With the knowledge the investigators have today, there is reason to believe that it is healthy to run both in a physical sense, but perhaps also in terms of brain function. However, there has not previously carried out extensive comparative studies of very active runners and healthy untrained control subjects. In this project the investigators will characterize the degree of training in subjects as the investigators will carry out various forms of physiological studies on the subjects' fitness level. The investigators will examine whether there is a linkage between training level and brain function.

The investigators will also examine muscle function at the molecular level. The investigators will isolate stem cells (satellite cells) from muscles biopsy and establish primary muscle cell cultures. By electrical stimulation of these cells in vitro, the investigators can emulate a muscle contraction as during physical activity. The investigators will test the overall hypothesis that physical activity affects stem cell function.

The investigators will further study whether epigenetic phenomena (methylation) of selected DNA sequences are sensitive to training level.

ELIGIBILITY:
Inclusion Criteria:

* 10 marathons, 2 within the last year or 50 km/week the last 5 years

Exclusion Criteria:

* smokers, any medication, chronic diseases, digestion of performance enhancing drugs, pregnancy, alcohol abuse

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Runners with high amount of training
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Fitness | one day
  Lactate threshold VO2max Running economy Lactate Peak
Cognitive Function | one day
  Memory, concentration, personality, intelligence
Blood | one day
  3 hour Oral Glucose Tolerance test (glucose, insulin, c-peptide) Fasting blood measurements ( lever, kidney, immune system, colesterol parameters) DNA
Muscle biopsy | one day
  Gene transcription Methylation
Body Composition | one day
  DXA scanning: Fat%, muscle mass, lean body mass, BMD MR scanning: Amount of visceral fat, volume of thighs

SECONDARY OUTCOMES:
Activity level and diet | 7 days
  Subjects are carrying a step pedometer for 7 days They are registrering their diet for 4 days They are answering questionaires about daily activity level and health now and in the past

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, Doctor, Study Director — Center of Inflammation and Metabolism
Locations (1):
- Center of Inflammation and Metabolism, Rigshospitalet, Copenhagen, Denmark